CLINICAL TRIAL: NCT03535935
Title: Efficacy, Safety and Response Predictors of Adjuvant Astragalus Therapy for Diabetic Kidney Disease (READY) - An Open-label Randomised Controlled Trial With Responder Regression Analysis
Brief Title: Efficacy, Safety and Response Predictors of Adjuvant Astragalus Therapy for Diabetic Kidney Disease
Acronym: READY
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: School of Chinese Medicine, The University of Hong Kong (Unknown)
Responsible Party: Principal Investigator, Sydney CW TANG, Chair of Renal Medicine and Yu Professor in Nephrology, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RE-02
Record Dates: First submitted 2018-05-13; First posted 2018-05-24 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Nephropathies; Diabetic Kidney Disease
Keywords: Chinese medicine; Astragalus; Pragmatic trial
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Huang Qi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessment of primary outcomes is performed by an independent laboratory
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard medical care (Active Comparator): Angiotensin converting enzyme inhibitor or angiotensin receptor blocker and oral hypoglycemic agents or insulin
  Interventions: Other: Routine medical care (active comparator)
- Add on astragalus powder (Experimental): 3 grams of water soluble astragalus sachets (equivalent to 15g raw herbs) administrated orally on top of standard medical care for 48 weeks.
  Interventions: Drug: Astragalus Powder; Other: Routine medical care (active comparator)

INTERVENTIONS:
Drug: Astragalus Powder — 3 grams of water soluble astragalus sachets (equivalent to 15g raw herbs) administrated orally on top of standard medical care for 48 weeks.
  Patients will have 5 days of medicine per week and will be advised to take the medicine once daily dissolved in boiling water in the first 5 days of the week.
  Arms: Add on astragalus powder
Other: Routine medical care (active comparator) — Angiotensin converting enzyme inhibitor or angiotensin receptor blocker

SUMMARY:
This add-on open-label randomised controlled pragmatic trial aims to:

1. evaluate the effect of add-on astragalus treatment on type 2 diabetic patients with stage 2 to 3 chronic kidney disease and macroalbuminuria.
2. estimate treatment effect, variance, recruitment rate, attrition rate and change in clinical manifestation including Chinese medicine syndrome for parameters optimisation and feasibility assessment for a subsequent phase III randomised controlled trial.
3. assess response predictors for efficacy and safety among type 2 diabetic patients with stage 2 to 3 chronic kidney disease and macroalbuminuria receiving add-on astragalus treatment

DETAILED DESCRIPTION:
This add-on open-label randomised controlled pragmatic trial.

Sample size is calculated based on planned regression analysis. We believe an annual GFR benefit of 5 ml/min/1.73m2 is deemed significant clinically. 118 patients are therefore needed to offer a power of 70% to detect a GFR difference of 5 ml/min/1.73m2 over 48-week allowing 15% attrition rate for this study with a significance level of alpha equals to 0.05.

A trial management committee (TMC) formed by PA, Co-As and RA will centralise all the data of the trial. Co-As and RA will collect, clean and send the data of patients to TMC on a weekly basis. All data will be double entered to computer and cleaned before analysis to prevent data entry errors. All data transfer will be encrypted to protect patients' confidentiality. TMC will have regular meetings monthly with experts to discuss the progress of the trial. An independent Data Monitoring Board (DMB) will be invited to monitor the progress of the trial. DMB will advise ethics committee to terminate the trial if data is showing extreme benefits or harm. Detailed guidelines will be discussed and set by DMB.

Missing values will be imputed with last observation carried forward. Patient without a postrandomisation assessment for a particular efficacy endpoint will be excluded from the analysis of that endpoint.

Regression analysis will be used to compare the adjusted mean of eGFR, UACR, HbA1c, FBG, and other biomarkers at week 48 between groups and statistical significance. The adverse events will be analysed in a narrative manner. The percentage of all adverse events and the rate of attrition due to adverse events will be compared between intervention groups and control groups.

To minimise Type I error inflation, the analysis will follow a hierarchical approach in the order of 1) comparison of baseline to end of treatment on eGFR and UACR; 2) comparison of baseline to end of treatment on other outcome measurements; 3) comparison of baseline to treatment midpoints on eGFR and UACR and 4) comparison of baseline to treatment midpoints on other outcome measurements.

Subgroup analysis will be performed for different age groups, gender chronic kidney disease stage and severity of albuminuria.

The dependent variable is the treatment response which is categorised into:

1. Improved or stabilised renal function, defined as eGFR after 48-week treatment being higher or equal to baseline.
2. Non-responder, defined as patients having eGFR decreased at a rate of less than 5 mL/min/1.73m2 after 48-week treatment compared to baseline.
3. Rapid deteriorating renal function, defined as eGFR of more than 5 mL/min/1.73m2 after 48-week treatment compared to baseline.

Potential prognostic variables (baseline values) include:

1. Demographics and past medical history: Age, gender, body mass index (BMI), systolic blood pressure, history and duration of smoking and alcohol consumption and others
2. Chinese medicine diagnosis: presence of Chinese medicine syndromes (e.g. spleen and kidney qi deficiency) based on the presentation of standardised and commonly documented signs and symptoms
3. Biochemical profile

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes for at least 5 years;
* with an estimated glomerular filtration rate (GFR) ≥30 ˂90 mL/min/1.73m2 confirmed with repeat testing over three or more months calculated by the abbreviated MDRD study equation;
* persistent macroalbuminuria with spot urine albumin-to-creatinine ratio (UACR) ≥ 300 mg/g confirmed by at least 2 out of 3 consecutive first morning void urine samples;
* on stable dose of anti-diabetic drug including insulin for 12 weeks;
* on stable dose of angiotensin-converting-enzyme inhibitor or angiotensin receptor blocker for 12 weeks; and
* willing and able to give written informed consent

Exclusion Criteria:

* with known history of glomerulonephritis, polycystic kidney disease, systemic lupus erythematosus, any suggestive evidence of nondiabetic glomerulopathy;
* with known history of kidney transplant;
* with concurrent severe disorders of heart, brain, liver, and hematopoietic system, tumor and mental disorder;
* with deranged liver function;
* poorly controlled blood pressure;
* with known history of intolerance or malabsorption of oral medications;
* with uncontrollable urinary infection;
* experiencing pregnancy; or
* participating in other clinical trial within 30 days

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in estimated GFR | From baseline to 48 weeks after treatment
  Efficacy and safety
Change in spot urine albumin-to-creatinine ratio | From baseline to 48 weeks after treatment
  Efficacy and safety

SECONDARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline to 48 weeks after treatment
Change in urinary monocyte chemotactic protein 1 (MCP-1) | From baseline to 48 weeks after treatment
Change in urinary Cystatin C | From baseline to 48 weeks after treatment
Change in lipids | From baseline to 48 weeks after treatment

OTHER OUTCOMES:
Change in biomarkers related to inflammation and fibrosis | From baseline to 48 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sydney CW TANG, MD, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - School of Chinese Medicine, Hong Kong

REFERENCES:
- [Derived] Chan KW, Kwong ASK, Tsui PN, Chan GCW, Choi WF, Yiu WH, Cheung SCY, Wong MMY, Zhang ZJ, Tan KCB, Lao L, Lai KN, Tang SCW; READY and SCHEMATIC research group. Add-on astragalus in type 2 diabetes and chronic kidney disease: A multi-center, assessor-blind, randomized controlled trial. Phytomedicine. 2024 Jul 25;130:155457. doi: 10.1016/j.phymed.2024.155457. Epub 2024 Feb 28. PMID 38810556
- [Derived] Chan KW, Kwong ASK, Tsui PN, Cheung SCY, Chan GCW, Choi WF, Yiu WH, Zhang Y, Wong MM, Zhang ZJ, Tan KCB, Lao L, Tang SCW. Efficacy, safety and response predictors of adjuvant astragalus for diabetic kidney disease (READY): study protocol of an add-on, assessor-blind, parallel, pragmatic randomised controlled trial. BMJ Open. 2021 Jan 12;11(1):e042686. doi: 10.1136/bmjopen-2020-042686. PMID 33436470